CLINICAL TRIAL: NCT03005626
Title: Transition From Adolescents to Adulthood for Patients With Congenital Patients With Congenital Heart Diseases: Impact of a Therapeutic Education Program on Quality of Life
Brief Title: Transition From Adolescents to Adulthood for Patients With Congenital Heart Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9752
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Congenital Heart Diseases
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic education (Experimental): Structured therapeutic education programs
  Interventions: Other: Therapeutic education
- Control group (Active Comparator): standard outpatient follow-up
  Interventions: Other: Standard follow-up

INTERVENTIONS:
Other: Therapeutic education
  Arms: Therapeutic education
Other: Standard follow-up
  Arms: Control group

SUMMARY:
The Investigators aim to measure the impact of a transition program in congenital cardiology in terms of health-related quality of life.

DETAILED DESCRIPTION:
The number of adults with congenital heart diseases (CHD) is increasing. However, many young adults are lost to follow-up even in experienced tertiary care centers. American and European guidelines recommend to improve the management of young adults with CHD. Structured therapeutic education programs are therefore needed to optimize the transfer to adult healthcare. Our tertiary care CHD center recently implemented a transition program and simultaneously investigators decided to measure its impact. Indeed investigators need data from randomized trials in this filed. After previous controlled quality of life studies among children and adults with CHD, investigators chose to use the health-related quality of life (HR-QoL) as primary endpoint in this randomized study to focus on patient related outcomes.

The investigators assume that patients who participate in this program will improve their quality of life compared to controls. If investigators demonstrate the benefit of this program, it will have important consequences for patients with CHD and eventually for patients with other chronic medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 13 years to 25 years inclusive.
* Carrying of Congenital Heart Disease as defined in the International Classification.
* Possible follow-up for one year on one of the three hospital center.
* Informed consent of the patient for adults and, parents or legal guardians for minors.
* Affiliation to a social security system.

Exclusion Criteria:

* Non-francophone,
* Severe intellectual impairment.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
PedsQL 4.0 score | Follow up of patients over 12 months
  Evolution of the quality of life assessed by PedsQL 4.0 self-reported scores from month 0 to month 12.

SECONDARY OUTCOMES:
Physiological parameters | Follow up of patients over 12 months
  Evolution of the physiological parameters during a cardiopulmonary exercise test performed on a treadmill according to a modified Bruce protocole. Evolution of the physiological parameters from month 0 to month 12
Ricci and Gagnon score | Follow up of patients over 12 months
  Evolution of the physical activity assessed by Ricci and Gagnon scores from month 0 to month 12. Ricci and Ganon score is a physical activity self-questionnaire with a total score out of 40 (<16 points: not very active, between 16 and 32 points: fairly active, > 32 points: very active).
Leuven Knowledge score | Follow up of patients over 12 months
  Evolution of the knowledge of the disease assessed by Leuven Knowledge scores from month 0 to month 12. The level of knowledge was assessed by the "transition readdiness assessment" instrument : 10-item questionnaire reflecting the basic knowledge of the diseases and its management.
Disease severity | Follow up of patients over 12 months
  The evolution of the severity of the disease from month 0 to month 12 was assessed by the degree of heart failure (NYHA functionnal class I to IV) and the number of hospitalizations (in stays and days) for complications related to the congenital heart disease
Anxiety and depression | Follow up of patients over 12 months
  The evolution of the levels of depression and/or anxiety from month 0 to month 12 was assessed respectively by :
  * the BDI (Beck Depression Inventory) for young adults
  * the CDI (Child Depression Inventory) for adolescents
  * the STAI (State and Trait Anxiety Inventory) for adults and STAI-C (Children) for adolescents.
  A higher score is associated with a higher risk of depression/anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

REFERENCES:
- [Result] Bredy C, Werner O, Huguet H, Guillaumont S, Auer A, Requirand A, Lavastre K, Abassi H, De La Villeon G, Vincenti M, Gavotto A, Vincent R, Pommier V, Dulac Y, Souletie N, Acar P, Karsenty C, Guitarte A, Berge M, Marguin G, Masseron MP, Pages L, Bourrel G, Engberink AO, Million E, Huby AC, Leobon B, Picot MC, Amedro P. Efficacy of a Transition Program in Adolescents and Young Adults With Congenital Heart Disease: The TRANSITION-CHD Randomized Controlled Trial. J Adolesc Health. 2024 Aug;75(2):358-367. doi: 10.1016/j.jadohealth.2024.04.022. Epub 2024 Jun 10. PMID 38864791
- [Derived] Werner O, Bredy C, Lavastre K, Guillaumont S, De La Villeon G, Vincenti M, Gerl C, Dulac Y, Souletie N, Acar P, Pages L, Picot MC, Bourrel G, Oude Engberink A, Million E, Abassi H, Amedro P. Impact of a transition education program on health-related quality of life in pediatric patients with congenital heart disease: study design for a randomised controlled trial. Health Qual Life Outcomes. 2021 Jan 19;19(1):23. doi: 10.1186/s12955-021-01668-1. PMID 33468144